CLINICAL TRIAL: NCT04759248
Title: A Phase II With 2 Parallel Cohorts Clinical Trial Targeting Estrogen Receptor Negative or PAM50 Non-luminal Disease With Atezolizumab in Combination With Trastuzumab and Vinorelbine in HER2-positive Advanced/Metastatic Breast Cancer - ATREZZO Study
Brief Title: Study With Atezolizumab in Combination With Trastuzumab and Vinorelbine in HER2-positive Advanced/Metastatic Breast Cancer
Acronym: ATREZZO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1907; 2020-000245-13 (EudraCT Number)
Record Dates: First submitted 2021-01-28; First posted 2021-02-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: cancer; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — atezolizumab; Trastuzumab; Vinorelbine

STUDY DESIGN:
Intervention Model Description: This is an open-label, single arm, Simon 2-stage, multicenter phase II study evaluating treatment with atezolizumab in combination with trastuzumab and vinorelbine in patients with locally advanced or metastatic PAM50 non-luminal/HER2+ BC refractory to trastuzumab based therapy and anti-HER2 ADC treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab in combination with Trastuzumab and Vinorelbine (Experimental)
  Interventions: Drug: Atezolizumab + Trastuzumab + Vinorelbine

INTERVENTIONS:
Drug: Atezolizumab + Trastuzumab + Vinorelbine — * Atezolizumab IV 1200 mg in combination with
  * Trastuzumab sc 600mg or IV 6mg/kg every 3 weeks and
  * Vinorelbine 25 mg/m² IV or 60 mg/m2 PO on days 1 and 8, every 3 weeks during the first cycle and if there are no toxicity signs dose will be increased to 80 mg/m2 PO o 30 mg/m2 IV.

SUMMARY:
Immune checkpoint inhibitors given in monotherapy in advanced breast cancer have shown modest benefit in first-line, but very limited efficacy in later lines. Thus, combination therapies are needed.

Response following anti-PD1/PD-L1 monotherapy is associated with large survival benefit in the advanced setting.

Previous studies of the intrinsic subtypes have shown that Basal-like and HER2-E are associated with higher expression of immune-related genes or higher infiltration of stromal tumor infiltrating lymphocytes compared to the luminal subtypes. Immune infiltration in BC is associated with chemo/antiHER2 responsiveness and potentially benefit from anti-PD-1/PD-L1 inhibitors.

In addition, one emerging biomarker of response to anti-PD-1 therapy is the tumor mutational burden (I.e. the total number of mutations per coding area of a tumor genome). The HER2-E and Basal-like profiles have been associated with high mutational burden.

A range of studies have been initiated including several phase II/III studies evaluating atezolizumab in combination with different chemotherapeutic compounds routinely used in breast cancer, but none with predefined biomarker beyond the expression of PD-L1 by IHC

ELIGIBILITY:
Inclusion Criteria:

* Male or female (Premenopausal or postmenopausal women)
* ECOG 0 to 2
* Histologically confirmed adenocarcinoma of the breast, metastatic or unresectable locally advanced.
* All patients must have received at least trastuzumab and other anti-HER2 ADCs (including but not limited to T-DM1).
* Measurable disease according to RECIST 1.1 criteria.
* Adequate organ function
* Baseline LVEF ≥50%
* Participants with asymptomatic brain metastases are eligible.

Exclusion Criteria:

* Treatment with any investigational anticancer drug within 14 days of the start of study treatment.
* Patient has received Vinorelbine or any other vinca alkaloids previously immediately prior to initiate study treatment.
* History of other malignant tumors in the past 3 years
* Known or suspected leptomeningeal disease (LMD)/ poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain metastases.
* Symptomatic hypercalcemia requiring treatment with bisphosphonates in the 14 days prior to inclusion
* Cardiopulmonary dysfunction
* Any other severe, uncontrolled
* Major surgery in the 28 days prior to enrolment
* Infection with HIV or active Hepatitis B and/or Hepatitis C.
* History of trastuzumab intolerance, including grade 3-4 infusion reaction or hypersensitivity.
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease,
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan. (Note: History of radiation pneumonitis in the radiation field [fibrosis] is permitted.)
* Active tuberculosis
* Receipt of a live, attenuated vaccine within 4 weeks prior to enrollment
* Prior treatment with CD137 agonists, anti-PD-1, or anti-PD-L1 therapeutic antibody or immune checkpoint targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug prior to enrolment
* Treatment with systemic immunosuppressive medications within 2 weeks prior to enrolment, or anticipated requirement for systemic immunosuppressive medications during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate | until disease progression or up to 2 years after treatment ends
  the proportion of patients with best overall response of complete response (CR) or partial response (PR), as per local investigator´s assessment and according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria

SECONDARY OUTCOMES:
Overall Response rate in PD-L1+ patients | until disease progression or up to 2 years after treatment ends
  the proportion of patients with best overall response of complete response (CR) or partial response (PR), as per local investigator´s assessment and according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
Clinical Benefit | 24 weeks
  Clinical Benefit Rate at 24 weeks
Overal survival | Until analysis data cutoff, 2 years
  Time from the date of allocation to the date of death due to any cause.
Progression free survival | 24 weeks
  Survival witouth observed progression
Duration of response | 24 weeks
  time from first documented response until progression
Time to response | 24 weeks
  time until first documented response
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | until end of treatment / through study completion, an average of 1 year
  AEs according to CTCAE v 5.0.
Overall Response rate in patients with brain metastases at baseline | Until disease progression or up to 2 years after treatment ends
  Patients with a history of brain metastases, current brain metastases, or equivocal brain lesions at baseline
Clinical Benefit in patients with brain metastases at baseline | 24 weeks
  Clinical Benefit Rate at 24 weeks in patients with a history of brain metastases, current brain metastases, or equivocal brain lesions at baseline
Progression free survival in patients with brain metastases at baseline | 24 weeks
  Survival without observed progression in patients with a history of brain metastases, current brain metastases, or equivocal brain lesions at baseline
Overal survival in patients with brain metastases at baseline | Until analysis data cutoff, 2 years
  Time from the date of allocation to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - H. Clínico San Cecilio de Granada, Granada, Andalusia
  - Hospital del Mar, Barcelona, Barcelona
  - Institut Català d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, La Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital de León, León
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No